CLINICAL TRIAL: NCT06803641
Title: The Effects of Mindfulness Practice With Tao Art (Love Peace Harmony Calligraphy and Song) on Well-being - Controlled Randomized Study
Brief Title: The Effects of Mindfulness Practice With Tao Art (Love Peace Harmony Calligraphy and Song) on Well-being
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sha Research Foundation (Other)
Responsible Party: Principal Investigator, Peter Hudoba De Badyn MD, FRCS, Principal Research Investigator, Sha Research Foundation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00083777
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Social Connectedness; Peace of Mind; Stress
Keywords: Well-being; Quality of life; Perceived Stress Scale; Social Connectedness Scale; Peace of Mind Scale; Randomization; Wait-list; Tao Calligraphy; Love Peace Harmony; Healing Art; Chinese Calligraphy

STUDY DESIGN:
Intervention Model Description: The study will be performed as a 6-month randomized wait-list control study. The participants will be adults (19 years and older). New participants may enter the study at any time and will be randomized into either the practice group or the wait-list control group.
  The practice group will start practices at the baseline zero time point and will stop their practices at the 3-months time point. The wait-list control group will crossover to the practice group at the three months time point and will stop practices at the 6-months time point.
  The study will evaluate the effects of mindfulness practice using these standardized questionnaires:
  * Perceived Stress Scale (PSS)
  * Social Connectedness Scale (SCS)
  * Peace of Mind Scale (PMS) All participants will complete the set of all three questionnaires upon entry into the study - the baseline zero time point; and again, at the 3-months and the 6-months time points.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practice Group (Experimental): The Practice group will start practices at baseline zero time point and will stop practices after three months at the 3-months time point. Participants in the Practice group will practice Mindfulness practice with Calligraphy at least 30 minutes daily for three months. All participants in the Practice group will complete the set of all three questionnaires upon entry into the study - at the baseline zero time point; at the 3-months time point and at the 6-months time point.
  Interventions: Other: Mindfulness practice with Tao Art (Calligraphy and Song Love Peace and Harmony).
- Wait-list Control Group (Other): The Wait-list Control group will crossover to become Practice group at the 3-months time point. Participants will start practices at the 3-months time point and will stop practices after three months at 6-months time point.
  All participants in Wait-list Group will complete the set of all three questionnaires upon entry into the study at baseline zero time point; at 3-months time-point and at 6-months time point.
  Interventions: Other: Mindfulness practice with Tao Art (Calligraphy and Song Love Peace and Harmony).

INTERVENTIONS:
Other: Mindfulness practice with Tao Art (Calligraphy and Song Love Peace and Harmony). — During mindfulness practice with Tao Art (Calligraphy and Song Love Peace Harmony), participants will repeatedly trace the lines of calligraphy with fingers while listening to, singing, or chanting with Tao Song. This enables them to achieve deep concentration, while maintaining fully alert state. The practice can be done in sitting or standing, depending on the health status and age and will last 30 minutes and is done daily for three months.

SUMMARY:
The Effects of Mindfulness Practice with Tao Art ("Love Peace Harmony" Calligraphy and Song) on Well-being - Controlled Randomized Study

The goal of this controlled randomized clinical study is to learn if a Tao Calligraphy Mindfulness Practice works to improve Well-being. The main questions it aims to answer are:

* Does Tao Calligraphy Mindfulness practice improve these three aspects of well-being in adults: (1) Perceived Stress, (2) the Social Connectedness, and (3) Peace of Mind?
* Will any improvement in the Perceived Stress Scale (PSS), the Social Connectedness Scale (SCS), and the Peace of Mind Scale (PMS) in adults be statistically significant? Investigators will compare the values of these three scales at the beginning of the mindfulness practices to their values at three months of practice and control groups.

Participants will:

* be randomized into practice and wait-list control groups
* complete the set of three questionnaires upon entry into the study - (the baseline or zero time point; at the 3-months time point, and at the six-months time point
* practice the mindfulness techniques with Tao Calligraphy and Tao Song for a minimum of thirty minutes daily

DETAILED DESCRIPTION:
Objective

The goal of this study is to measure the positive effects of a unique form of mindfulness practice that involves engaging with Tao art (tracing the Tao Calligraphy "Love Peace Harmony" while listening to or singing the Tao Music or Tao Song "Love, Peace and Harmony") on human adult well-being. Investigators will study the impact of this Tao art mindfulness practice on three aspects of well-being: Perceived Stress, Social Connectedness and Peace of Mind.

Hypotheses

The research null hypothesis is that participants who will engage in daily mindfulness practice with Tao art will report NO significant improvement in three aspects of well-being as measured by standardized scientific questionnaires; specifically, NO significant reduction of Perceived Stress, NO significant increase in Social Connectedness and NO significant increase in Peace of Mind.

For statistical analysis of scores obtained from questionnaires, the Anova and regression analysis will be used to evaluate the null hypothesis. The p value will represent how unlikely the observed data would be if the null hypothesis were actually true and investigators will use them to reach conclusions. The confidence level is set at 95% and if we receive p < 0.05, then H0 is rejected. The correlation coefficient will be used to determine any correlation between various factors (e.g. effects of age, sex, length, and frequency of mindfulness practices and other) on outcome and regression analysis will be used to determine the relation of independent and dependent variables.

Background and Theoretical Framework

Human interest in "well-being" dates back thousands of years, from complex indigenous understandings through to the ancient Greeks. However, a clear and useful definition and conceptualization of well-being remains elusive, a situation which has manifested historically, contemporarily, to the public, and within and across disciplines.

The investigators concur more with Lomas and VanderWeele's understanding of well-being as related to health and flourishing and Joshanloo's focus on mental balance, defined as a sense of tranquility resulting from inner peace and harmonious interactions with the external environment, and life satisfaction.

A large and growing body of research shows that mindfulness and meditation practices are beneficial to physical and mental health and well-being. Mindfulness refers to a state of awareness that arises from paying attention to the present moment, without judgment, whereas meditation refers to a practice or technique that can cultivate mindfulness, inner peace, and more. Mindfulness practices are often synonymous with meditation, and the terms are often used interchangeably.

Research has demonstrated the positive effects of mindfulness-based meditation on brain function, immune system function, diabetes, hypertension, fibromyalgia, cholesterol levels, blood pressure, heart rate, and cortisol levels. Likewise, mindfulness and meditation practices have been shown to increase self-compassion and improve memory and emotional regulation. In a comprehensive meta-analysis of 209 studies, the authors concluded that mindfulness-based therapy was effective for many types of psychological problems, while being especially good for reducing anxiety, depression, and stress. In another overall review of mindfulness-based interventions, they were found to be effective for many common and diverse mental, physical, and social conditions.

In recent decades, mindfulness and meditation practices and programs have become increasingly commonplace for stress management and reduction because they are effective. It is no wonder that mindfulness-based meditation practices lead to greater mental, physical, and psychological well-being, with one of the key mechanisms for such outcomes being their effect on the regulation or reduction of stress.

Besides mindfulness and meditation practices, the interest in the application of the arts for public health and well-being has also grown in recent years. Self-expression through art or engaging with different forms of art has been found to be helpful for many health conditions, and doctors in the United Kingdom have started prescribing "the arts" to treat or positively influence many kinds of health conditions.

Some forms of art are also meditative and contemplative, and many can be readily transformed into such a process. The mindfulness-based meditation being explored in this research rests in part on the benefits of music, singing or chanting, and calligraphy tracing (in particular, tracing a unique form of Chinese calligraphy).

Through the personal experiences, everyone knows that music can transform or uplift the mood and research supports this, suggesting that engagement with music plays a role in mood regulation. Harvard Health shares how music enhances our health and performance, claiming that music has "major effects on many aspects of health, ranging from memory and mood to cardiovascular function and athletic performance." A recent systematic review and meta-analysis of "music interventions" found that they are associated with significant clinical improvements in Health-Related Quality of Life indices (especially the mental components) and, interestingly, they found that whether people sang, played, or listened to music, the results were similar. A slightly earlier systematic review and meta-analysis of music therapy for stress reduction found overall large to medium-large effects on stress-related outcomes. Likewise, though research is limited in this area, chanting meditations have documented effects on stress and well-being.

Chinese calligraphic writing is a dynamic process that uses an ink-laden brush to create defined configurations of characters. Revered as one of the most important art forms in China, as a mindfulness practice, it has also been shown to help reduce stress and improve mental well-being. The practice of Chinese calligraphy writing facilitates the development of concentration, creativity, and relaxation, which can lead to a more peaceful mental state. Studies in the medical field have confirmed its significant effects on psychosomatic conditions, post-traumatic hyper-arousal symptoms, hypertension, and type 2 diabetes. Other research publications have shown how it can improve cognitive function in the elderly, improve neuropsychiatric symptoms, and reduce stress. In one case, a man who was in a coma for two years awakened and continued to improve after his medical team took his hand and helped him to trace calligraphy daily with his finger.

This research will explore the effects of a unique mindfulness-based meditation that combines tracing the Tao Calligraphy "Love Peace Harmony" while listening to, singing, or chanting the Tao Song "Love, Peace and Harmony." Investigators will study its effect upon selected aspects of well-being.

Tao Calligraphy is based on a unique branch of Chinese calligraphy known as Yi Bi Zi, which applies one-stroke writing. Every character is written with one continuous stroke of the brush, with the brush always in contact with the paper.

In a unique style of moving meditation, participants will focus on a work of Tao Calligraphy art, tracing the characters with their fingers while simultaneously listening to or singing/chanting (silently or aloud) the Tao Music or Song, which enables them to achieve deep concentration and relaxation during wakefulness.

The Tao Song "Love, Peace and Harmony" consists of short, inspiring verses that are repeated, and is a beautiful way to lift and inspire peoples' hearts and help them to experience peace and calm. The song was professionally recorded and is available on the Love Peace Harmony Foundation's website as a free distribution.

The investigators have already discussed the value of Tao art mindfulness meditations for improving depression, anxiety, pain, and health, and how this appears to contribute to numerous beneficial outcomes related to well-being by the Short Form 36-item (SF-36) questionnaire to measure quality of life and by the European Organization for Research and Treatment of Cancer 30-item core quality of life questionnaire (EORTC QLQ C-30). In this study, the investigators will measure other aspects of well-being, namely perceived stress, peace of mind, and social connectedness.

ELIGIBILITY:
Inclusion criteria

* Age 19 and over
* Willingness and ability to comply with data collection requirements
* Submission of required documentation before entering the study, including informed consent and consent to release of information
* Willingness to allow their data to be used for research purposes and published as deemed fit (while conforming to all applicable privacy laws) by Sha Research Foundation
* Willingness to practice the daily mindfulness practices for at least 30 minutes and follow the study protocol

Exclusion criteria

* Not meeting any of the inclusion criteria
* Unwillingness to participate in data gathering
* Unable to follow the practice regimen, including the daily individual mindfulness practices for at least 30 minutes
* Pregnant or nursing. Participants who become pregnant during the study will be required to end their participation.
* Serious mental disorders (e.g., schizophrenia)
* There is no exclusion criteria placed upon potential subjects related to national origin, culture, ethnicity, race, sex, physical disability, sexual orientation, religion, or spiritual practices.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-05 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Perceived Stress Scores on Perceived Stress Scale at three months | From start of Mindfulness practices with Tao Art (Calligraphy and Song Love Peace and Harmony) to end of practices at three months.
  The Perceived Stress Scale (PSS) measures the degree to which situations in one's life are appraised as stressful, will be used to assess the impact of the Tao art mindfulness practice on psychological stress.
  The PSS has ten scores derived from answers to the then questions of PSS. These ten scores have a 0-to-4 scale, with 4 being the best possible outcome. PSS score is determined by following these directions:
  First, investigators will reverse the scores for questions 4, 5, 7, and 8. On these four questions investigators will change the scores as follows: 0 to 4, 1 to 3, 2 to 2, 3 to 1, 4 to 0.
  Then, investigators will add up the scores for each item to get a total. Individual scores on the PSS can range from 0 to 40, with higher scores indicating higher perceived stress:
  * Scores ranging from 0-13 would be considered low stress.
  * Scores ranging from 14-26 would be considered moderate stress.
  * Scores ranging from 27-40 would be considered high perceived stress.
Mean Change from Baseline in Social Connectedness Scores on Social Connectedness Scale at three months | Frame: From start of Mindfulness practices with Tao Art (Calligraphy and Song Love Peace and Harmony) to the end of practices at three months.
  The Social Connectedness Score (SCS) measures the extent to which one feels connected to others in their social environment. It is derived from answers to eight questions along a 1-to-6 scale, 6 being the best possible outcome. The items are summed, with a higher total score indicating more connectedness to others.
Mean Change from Baseline in Peace of Mind Scores on Peace of Mind Scale at three months | Frame: From start of Mindfulness practices with Tao Art (Calligraphy and Song Love Peace and Harmony) to end of practices at three months.
  The Peace of Mind Scale (PMS) was developed to capture an internal state of peacefulness and harmony that is said to be a more valued aspect of subjective well-being in the east, however it has recently begun to receive attention cross-culturally and has also been studied in conjunction with calligraphy writing and stress.
  PMS has seven scores, derived from answers to the seven questions of PMS. These seven scores have a 1-to-5 scale, with 5 being the best possible outcome. PMS score is determined by following these directions:
  First, investigators will reverse the scores for questions 5 and 7. On these two questions investigators will change the scores as follows: 1 to 5, 2 to 4, 3 to 3, 4 to 2, 5 to 1.
  Then, investigators will add up the scores for each item to get a total. The average of the item scores is an overall measure of peace of mind, with higher scores indicating greater peace of mind.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hudoba De Badyn, MD, FRCS, Principal Investigator — Sha Research Foundation; Marsha Valutis, PhD, Principal Investigator — Sha Research Foundation
Locations (1):
- Private practice (Psychology), Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share the protocol with the statistical analysis plan of the study, the mean change from baseline in Perceived Stress Scores, Social Connectedness Scores, and in the Peace of Mind Scores after three months of mindfulness practices with Tao Art.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The protocol with the statistical analysis plan of the study will be available from February 28, 2025 until the end of the study on December 31, 2030.
  The mean change from baseline in Perceived Stress Scores, Social Connectedness Scores, and in the Peace of Mind Scores after three months of mindfulness practices with Tao Art will be available from December 31, 2030 until December 31, 2031.
Access Criteria: Anyone with an active account at this platform.

REFERENCES:
- [Result] Kao H Sr, Zhu L, Chao AA, Chen HY, Liu IC, Zhang M. Calligraphy and meditation for stress reduction: an experimental comparison. Psychol Res Behav Manag. 2014 Feb 13;7:47-52. doi: 10.2147/PRBM.S55743. eCollection 2014. PMID 24611024
- [Result] Pan A, Okereke OI, Sun Q, Logroscino G, Manson JE, Willett WC, Ascherio A, Hu FB, Rexrode KM. Depression and incident stroke in women. Stroke. 2011 Oct;42(10):2770-5. doi: 10.1161/STROKEAHA.111.617043. Epub 2011 Aug 11. PMID 21836097
- [Result] Kobau R, Seligman ME, Peterson C, Diener E, Zack MM, Chapman D, Thompson W. Mental health promotion in public health: perspectives and strategies from positive psychology. Am J Public Health. 2011 Aug;101(8):e1-9. doi: 10.2105/AJPH.2010.300083. Epub 2011 Jun 16. PMID 21680918
- [Result] White JD. National Cancer Institute's support of research to further integrative oncology practice. J Natl Cancer Inst Monogr. 2014 Nov;2014(50):286-7. doi: 10.1093/jncimonographs/lgu036. No abstract available. PMID 25749590
- [Result] Marikar Bawa FL, Mercer SW, Sutton JW, Bond CM. Mindfulness for people with chronic pain: Factors affecting engagement and suggestions for programme optimisation. Health Expect. 2023 Jun;26(3):1287-1307. doi: 10.1111/hex.13745. Epub 2023 Mar 12. PMID 36908018
- [Result] Jamil A, Gutlapalli SD, Ali M, Oble MJP, Sonia SN, George S, Shahi SR, Ali Z, Abaza A, Mohammed L. Meditation and Its Mental and Physical Health Benefits in 2023. Cureus. 2023 Jun 19;15(6):e40650. doi: 10.7759/cureus.40650. eCollection 2023 Jun. PMID 37476142
- [Result] Pascoe MC, de Manincor M, Tseberja J, Hallgren M, Baldwin PA, Parker AG. Psychobiological mechanisms underlying the mood benefits of meditation: A narrative review. Compr Psychoneuroendocrinol. 2021 Mar 10;6:100037. doi: 10.1016/j.cpnec.2021.100037. eCollection 2021 May. PMID 35757358
- [Result] Poissant H, Mendrek A, Talbot N, Khoury B, Nolan J. Behavioral and Cognitive Impacts of Mindfulness-Based Interventions on Adults with Attention-Deficit Hyperactivity Disorder: A Systematic Review. Behav Neurol. 2019 Apr 4;2019:5682050. doi: 10.1155/2019/5682050. eCollection 2019. PMID 31093302
- [Result] de Witte M, Orkibi H, Zarate R, Karkou V, Sajnani N, Malhotra B, Ho RTH, Kaimal G, Baker FA, Koch SC. From Therapeutic Factors to Mechanisms of Change in the Creative Arts Therapies: A Scoping Review. Front Psychol. 2021 Jul 15;12:678397. doi: 10.3389/fpsyg.2021.678397. eCollection 2021. PMID 34366998
- [Result] de Witte M, Lindelauf E, Moonen X, Stams GJ, van Hooren S. Music Therapy Interventions for Stress Reduction in Adults With Mild Intellectual Disabilities: Perspectives From Clinical Practice. Front Psychol. 2020 Dec 10;11:572549. doi: 10.3389/fpsyg.2020.572549. eCollection 2020. PMID 33362637

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT06803641/Prot_SAP_000.pdf